CLINICAL TRIAL: NCT02887651
Title: Cavity Boost Radiation Therapy vs. Observation in Cerebral Metastases After Complete Surgical Resection
Acronym: C-O-MET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5405
Record Dates: First submitted 2016-07-14; First posted 2016-09-02 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Metastases; Surgery
Keywords: cerebrale metastases; radiotherapy; surgery; complete surgical resection; resection; cavity boost radiation therapy; observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observation (No Intervention): patients in the observation arm receive no adjuvant local radiation therapy after complete surgical resection of a cerebral metastasis
- cavity boost radiation therapy (Active Comparator): patients in the intervention arm receive an adjuvant local radiation therapy (cavity boost radiation therapy: 10 x 3 Gy ad 30 Gy; clinical target volume (CTV): resection cavity plus surrounding 5 mm; planning target volume (PTV): CTV + 1mm)
  Interventions: Radiation: Cavity boost radiation

INTERVENTIONS:
Radiation: Cavity boost radiation — Cavity boost radiation therapy with 10 x 3 Gy for patients suffering from complete resected cerebral metastases
  Arms: cavity boost radiation therapy

SUMMARY:
The purpose of this study is to determine whether a local fractionated radiation therapy achieves a better local tumor control after complete surgical metastases resection at 6 month as compared to observation alone. Further it should be evaluated if cognitive functioning and quality of life is similar in both groups.

DETAILED DESCRIPTION:
The surgical resection of cerebral metastases as a key element in a multimodal therapeutic concept of brain metastatic patients is included in the common recommendations and international guidelines (level I evidence). These recommendations are based on a series of prospective, randomized and controlled studies which addressed the impact of the surgical metastases resection combined with a whole-brain radiation therapy (WBRT) in comparison to WBRT alone. Achieving local tumor control is the major goal of surgery and local tumor control rate after surgery alone has been addressed in few studies: A prospective, randomized American multicenter study revealed a local recurrence rate of 46% by median follow-up of 43 weeks for patients who underwent surgery alone without an adjuvant radiation therapy. Similarly, the 2-year local recurrence rate after metastases resection alone was 53.1% in a retrospective Korean study and 59% in the prospective, randomized and controlled EORTC 22952-26001 study.

In conclusion, standard surgery alone is not sufficient to achieve local control in about 50% of patients (evidence level I). Therefore, surgery of cerebral metastases is often followed by an adjuvant radiation therapy, which is an important part of a multi-modal therapy. Evidence for an additional adjuvant whole-brain radiation therapy (WBRT) after surgical resection was gained from a first prospective, randomized study in 1998: Patients treated by surgery followed by adjuvant WBRT had a significant lower local in-brain progression rate as compared to patients randomized to surgery alone (46% with a median follow-up of 48 weeks in the observation group vs. 10% with a median follow-up of 43 weeks). This result was recently confirmed by the EORTC 22952-26001 study: The 2-year local in-brain progression rate after surgical resection was reduced by a WBRT from 59% to 27%. But despite the lower local and also lower distant in-brain progression rate, the WBRT had no significant influence on the overall survival. The additional analysis of the quality of life data of the EORTC 22952-26001 study showed, that a WBRT negatively impacts the health-related quality of life with a statistically relevant and clinically significant impairment of the physical functioning (at 8 weeks), cognitive functioning and of the global health status. In conclusion, WBRT after surgery of cerebral metastases significantly reduces the incidence of local recurrences but has no impact on the overall survival and has a significant negative impact on the patient´s quality of life and cognitive function. Therefore, WBRT is not mandatory as adjuvant concept after surgical metastases resection and does not have an additional oncological impact in comparison to observation.

A local fractionated radiation therapy in analogy to the WBRT might achieve a similar local tumor control than observation alone but might be associated with an improved cognitive functioning as compared to WBRT. The purpose of this study is to determine whether a local fractionated radiation therapy achieves a better local tumor control after complete surgical metastases resection at 6 month as compared to observation alone. Further it should be evaluated if cognitive functioning and quality of life is similar in both groups.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastasis of carcinoma (except small cell carcinoma) or malignant melanoma
* 1-3 metastases in the preoperative MRI
* Karnofsky Performance Status (KPS) ≥ 70
* Age > / = 18 years
* Recursive partitioning analysis (RPA) 1-2
* life expectation ≥ 6 months
* no previous irradiation of the brain
* MRI examinations possible
* start of the radiation therapy possible within 6 weeks after surgery
* informed consent

Exclusion Criteria:

* confirmation of residual tumor in the postoperative MRI
* dementia or disease of central nervous system with a higher risk or radiogenic toxicity
* contraindication for MRIs or lack of acceptance for a MRI
* Glasgow Coma Scale < 12
* Severe concomitant disease: severe cardiac, pulmonary, renal diseases with an increased risk of surgery and radiation
* previous therapeutic irradiation of the brain
* no histological confirmation of carcinoma metastases or malignant melanoma metastases
* cerebral metastases of small cell cancer, undifferentiate neuro-endocrine carcinoma, lymphoma, leucemia, sarcoma or germ cell tumor
* leptomeningeal carcinosis
* distance of the cerebral metastasis to the optic system or radiation sensible brain parts < 10 mm
* metastases of the brain stem, Di- or Mesencephalons, Pons oder Medulla oblongata
* bone marrow dysfunction
* contrast agent allergy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Local tumor control of resected metastases at 6 month | 6 month
  Primary outcome measure is the local tumor control of resected metastases after local cavity boost radiation therapy or observation at 6 month

SECONDARY OUTCOMES:
Local tumor control of resected metastases at 12 and 18 month | 12, 18 month
  Secondary outcome measure is the local tumor control of resected metastases after local cavity boost radiation therapy or observation at 12 and 18 month
Distant tumor control of resected metastases at 6, 12 and 18 month | 6, 12 and 18 month
  Secondary outcome measure is the distant tumor control at 6, 12 and 18 month
Incidence of leptomeningeal carcinosis | 6, 12 and 18 month
  Secondary outcome measure is the incidence of a leptomeningeal carcinosis at 6, 12 and 18 month
Eortc qlq bn20 questionaire | 3, 6, 9 12, 15, 18 month
  Secondary outcome measure is the patients quality of life at 3, 6, 9 12, 15, 18 month as assessed by the Eortc qlq bn20 questionaire
Eortc qlq c30 questionaire | 3, 6, 9, 12, 15, 18 month
  Secondary outcome measure is the patients quality of life at 3, 6, 9, 12, 15 and 18 month as assessed by the Eortc qlq c30 questionaire
Mini-Mental State Examination (MMSE) | 3, 6, 9 12, 15, 18 month
  Secondary outcome measure is the patients neurocognitive functioning at 3, 6, 9 12, 15 and 18 month as assessed by the MMSE
Hopkins Verbal Learning Test (HVLT) | 3, 6, 9 12, 15, 18 month
  Secondary outcome measure is the patients neurocognitive functioning at 3, 6, 9, 12, 15 and 18 month as assessed by the Hopkins Verbal Learning Test (HVLT),
Controlled Oral Word Association (COWA) | 3, 6, 9 12, 15, 18 month
  Secondary outcome measure is the patients neurocognitive functioning at 3, 6, 9 12, 15 and 18 month as assessed by the Controlled Oral Word Association (COWA)
Test and Trail-Making Test (TMT) A & B | 3, 6, 9 12, 15, 18 month
  Secondary outcome measure is the patients neurocognitive functioning at 3, 6, 9 12, 15 and 18 month as assessed by the Test and Trail-Making Test (TMT) A & B

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sabel, Prof. Dr., Principal Investigator — Department of Neurosurgery; Wilfried Budach, Prof. Dr., Principal Investigator — department of radiation oncology
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided